CLINICAL TRIAL: NCT04339439
Title: Does Addition of a Vessel Loop in Wound Closure Improve Suture Removal?
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: A preliminary analysis was performed in this study halfway through enrollment and significant results were found, therefore the study was stopped.
Sponsor: Carilion Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-20-737
Record Dates: First submitted 2020-04-06; First posted 2020-04-09 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Patient Satisfaction; Suture, Complication
Keywords: suture; vessel loop; suture removal; satisfaction; carpal tunnel release
MeSH Terms: conditions — Patient Satisfaction; Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: Patients who agree to participate will be enrolled and randomized to one of two study groups:
  * Group 1: Incision closure without a vessel loop.
  * Group 2: Incision closure with a vessel loop.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Closure without vessel loop (No Intervention): These patients will receive standard of care closure of the carpal tunnel release incision.
- Closure with vessel loop (Experimental): These patients will receive closure of the carpal tunnel release incision with a vessel loop placed under the sutures.
  Interventions: Device: Vessel loop (FDA product code FZZ)

INTERVENTIONS:
Device: Vessel loop (FDA product code FZZ) — The intervention will be a vessel loop placed below sutures to raise the sutures from the skin of the palm.
  Arms: Closure with vessel loop

SUMMARY:
This study will investigate whether adding a vessel loop under sutures after elective carpal tunnel release increases patient satisfaction with suture removal.

DETAILED DESCRIPTION:
Surgical wound closure with nonabsorbable stitches necessitates subsequent suture removal, a process that can be uncomfortable for the patient and consume clinic time and resources. Anecdotal evidence suggests that the addition of a vessel loop under the sutures both simplifies suture removal and reduces discomfort. In this study, we propose a prospective, randomized, controlled, superiority trial to assess the impact of a vessel loop wound closure and suture removal for elective carpal tunnel release (CTR). Patients will be prospectively enrolled to one of two groups: closure without a vessel loop or closure with a vessel loop. The primary outcome measure will be patient satisfaction with suture removal. Time for wound closure, time for suture removal, pain with suture removal and other patient reported outcomes will be measured. These data will allow us to determine the benefit of addition of a vessel loop in wound closure.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective primary CTR (CPT 64721) at Carilion Clinic for carpal tunnel syndrome (CTS) diagnosed by CTS-6 or electrodiagnostic studies (EDS).

Exclusion Criteria:

* Emergency procedures.
* Revision procedures.
* Bilateral procedures.
* Concomitant procedures.
* Inability to provide informed consent for the study.
* Non-native English speakers.
* Allergy to suture material.
* History of wrist trauma.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-11-23 (Actual); Study Completion 2022-07-19 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction with suture removal | First postoperative visit (1-2 weeks)
  This will be measured on a 100mm visual analog scale.

SECONDARY OUTCOMES:
Pain with suture removal | First postoperative visit (1-2 weeks).
  This will be measured on a 100mm visual analog scale.
Time to close the surgical wound | Intraoperatively (0 days)
  The time that it takes the provider to close the wound intraoperatively.
Time to remove suture | First postoperative visit (1-2 weeks).
  The time that it takes the provider to remove sutures postoperatively.
Wound complications | 6 weeks postoperatively
  Any wound complications will be noted from the clinical record.
QuickDASH | 6 weeks postoperatively.
  A validate instrument assessing disability of the arm, shoulder, and hand.

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Apel, MD, PhD, Principal Investigator — Carilion Clinic
Locations (1):
- Carilion Institute for Orthopaedics & Neurosciences, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
No IPD are to be shared with other researchers. Only aggregate data will be shared.